CLINICAL TRIAL: NCT00755495
Title: A Phase 2, Double-Blind, Randomized, Placebo-Controlled, Parallel-Group, Multicenter Proof-of-Concept Study to Evaluate the Safety and Efficacy of Ramelteon Taken in Combination With Doxepin for the Treatment of Subjects With Chronic Insomnia
Brief Title: Safety and Efficacy of Ramelteon and Doxepin in Subjects With Chronic Insomnia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-05-TL-375-067; U1111-1114-2536 (Registry Identifier: WHO)
Record Dates: First submitted 2008-09-17; First posted 2008-09-19 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: Chronic Insomnia; DIMS (Disorders of Initiating and Maintaining Sleep); Disorders of Initiating and Maintaining Sleep; Insomnia Disorder Sleep Initiation Dysfunction; Transient Insomnia; Drug Therapy; Sleep Disorders, Intrinsic
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Disorders, Intrinsic | interventions — ramelteon; Doxepin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Ramelteon 8 mg QD and Doxepin 3 mg QD (Experimental)
  Interventions: Drug: Ramelteon and doxepin
- Ramelteon 8 mg QD and Doxepin Placebo QD (Experimental)
  Interventions: Drug: Ramelteon
- Ramelteon Placebo QD and Doxepin 3 mg QD (Active Comparator)
  Interventions: Drug: Doxepin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ramelteon and doxepin — Ramelteon 8 mg, tablets, orally, once daily and doxepin 3 mg, liquid, orally, once daily for up to five weeks.
  Other Names: Rozerem™; TAK-375; Sinequan®; ramelteon
  Arms: Ramelteon 8 mg QD and Doxepin 3 mg QD
Drug: Ramelteon — Ramelteon 8 mg, tablets, orally, once daily and doxepin placebo-matching liquid, orally, once daily for up to five weeks.
  Other Names: Rozerem™; TAK-375
  Arms: Ramelteon 8 mg QD and Doxepin Placebo QD
Drug: Doxepin — Ramelteon placebo-matching tablets, orally, once daily and doxepin 3 mg, liquid, orally, once daily for up to five weeks.
  Other Names: Sinequan®
  Arms: Ramelteon Placebo QD and Doxepin 3 mg QD
Drug: Placebo — Ramelteon placebo-matching tablets, orally, once daily and doxepin placebo-matching liquid, orally, once daily for up to five weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy of ramelteon, once daily (QD), combined with doxepin in treating subjects with insomnia.

DETAILED DESCRIPTION:
Approximately 60 to 70 million adults in the United States alone are affected by insomnia. Daytime symptoms of insomnia include tiredness, lack of energy, difficulty concentrating, and irritability. Recent epidemiologic research focusing on quality of life has identified significant insomnia-related morbidities that relate to work productivity, health care utilization, and risk of depression. Insomnia is also associated with diminished work output, absenteeism, and greater rates of accidents. Gamma-aminobutyric acid is the major inhibitory transmitter in the central nervous system and most currently prescribed sleep agents are benzodiazepine receptor agonists, which induce sleep by binding to the benzodiazepine receptor site of the gamma-aminobutyric acid -A receptor complex. In addition to sleep, benzodiazepine receptor agonists can cause a wide range of ancillary effects not directly related to sleep, including sedative, anxiolytic, muscle-relaxant, and amnesic effects, and have risks of tolerance, dependence, and abuse potential.

Doxepin is one of a class of psychotherapeutic agents known as dibenzoxepin tricyclic compounds. Doxepin is indicated for the treatment of depression, anxiety, and psychotic depressive disorders. The most common adverse event associated with the use of doxepin is drowsiness. A limited number of controlled studies have been performed to examine the effects of low doxepin on insomnia.

TAK-375 (Ramelteon) is a melatonin receptor agonist with affinity for the human melatonin receptor subtype 1 (MT1), melatonin receptor subtype 2 (MT2) and selectivity over the melatonin receptor subtype 3 (MT3) receptor.

This trial will determine if the co-administration of ramelteon and doxepin will decrease both latency to persistent sleep and wake time after sleep onset. Study participation is anticipated to be about 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Based on sleep history, the subject has had primary insomnia as defined by the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition Revised (DSM-IV-TR™) for at least 3 months.
* Female patients of childbearing potential must be nonpregnant and nonlactating, and utilizing an acceptable method of contraception.
* Has a body mass index between 18 and 34 inclusive (weight/height2).
* Based on sleep history, the subject reports subjective sleep latency greater than or equal to 45 minutes and reports wake time after persistent sleep onset of greater than or equal to 45 minutes.
* The subject has an average wake time after persistent sleep onset of at least 60 minutes as determined by polysomnography during Screening (Day -7 PM through Day -5 AM). Wake time after persistent sleep onset must be greater than or equal to 30 minutes each night of polysomnography Screening.
* In addition to meeting the criteria for wake time after persistent sleep onset, must have an average latency to persistent sleep of at least 20 minutes as determined by polysomnography during Screening (Day -7 PM through Day -5 AM). Latency to persistent sleep must be greater than or equal to 15 minutes each night of polysomnography Screening.
* Based on sleep history, the subject's habitual bedtime is between 9:00 PM and 1:00 AM.
* Is willing to have a fixed bedtime and agrees to go to bed within +/-30 minutes of the habitual bedtime during the entire study.
* Is willing to remain in bed for at least 8 hours each night during the entire study.
* Based on sleep history, the subject either has not been using pharmacological assistance to sleep or uses pharmacological assistance no more than 4 times per week during the 3 months prior to Initial Screening. Subjects must agree to discontinue the use of all pharmacological sleep aids beginning 1 week prior to polysomnography Screening and throughout the entire duration of the study.
* Has consistent access to a touch-tone phone and are willing to complete telephone questionnaires during participation in the study.

Exclusion Criteria:

* Has a known hypersensitivity to doxepin or related compounds (tricyclic antidepressants), or ramelteon or related compounds, including melatonin, and 5-hydroxytryptophan.
* Has participated in any other investigational study and/or taken any investigational drug within 30 days prior to the first dose of single-blind study medication.
* Has sleep schedule changes required by employment (eg, shift worker) within 3 months prior to the first dose of single-blind study medication.
* Has flown across greater than 3 time zones within 7 days prior to Initial Screening, or will travel across 2 or more time zones during the course of the study.
* Has participated in a weight loss program or has substantially altered their exercise routine within 30 days prior to the first dose of single-blind study medication.
* Is required to take or intends to continue taking any disallowed medication or any prescription medication or over-the counter medication that is known to affect the sleep/wake function or otherwise interfere with evaluation of the study medication, including:

  * Anxiolytics central nervous system active drugs (including herbal).
  * Hypnotics Narcotic analgesics.
  * Antidepressants Beta blockers.
  * Anticonvulsants St. John's Wort.
  * Sedating H1 antihistamines Kava-kava.
  * Systemic steroids Ginkgo-biloba.
  * Respiratory stimulants over-the-counter and prescription stimulants.
  * Sedating decongestants over-the-counter and prescription diet aids.
  * Antipsychotics over-the-counter sleep aids.
  * Muscle relaxants.
  * Melatonin and all other drugs or supplements known to affect sleep/wake function.
* Has ever had a history of fibromyalgia, glaucoma, seizures (excluding childhood febrile seizures), sleep apnea, and/or chronic obstructive pulmonary disease.
* Currently has, or has had a diagnosed history of psychiatric disorder as defined in DSM-IV-TR™ (including anxiety, depression, suicidal ideation, mental retardation, cognitive disorder, bipolar illness and schizophrenia) within the past 6 months of Initial Screening.
* Has a history of drug addiction or drug abuse as defined in DSM-IV-TR™ within the past 12 months of Initial Screening.
* Has a history of alcohol abuse within the past 12 months, as defined in DSM-IV-TR™ and/or regularly consumes more than 2 alcoholic drinks per day.
* Has a current significant hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, hematological, metabolic or neurological disorders, or tendency for urinary retention, unless currently controlled and stable with protocol-allowed medication, within 30 days prior to the first dose of single-blind study medication.
* Has a previous history of cancer, other than basal cell carcinoma, that has not been in remission for at least 5 years prior to the first dose of single-blind study drug. (This criterion does not apply to subjects with basal cell or Stage 1 squamous cell carcinoma of the skin).
* Uses tobacco products or any other products that may interfere with the sleep wake cycle during nightly awakenings.
* Has used any central nervous system medication or other drugs or supplements known to affect sleep/wake function within 1 week (or 5 half lives of the drug, whichever is longer) prior to the administration of single-blind study medication. These medications must not have been used to treat psychiatric disorders.
* Has used melatonin, or other drugs or supplements known to affect sleep/wake function within 1 week (or 5 half lives of the drug, whichever is longer) prior to the first dose of single-blind study medication.
* Has any clinically important abnormal finding as determined by a medical history, physical examination, electrocardiogram, or clinical laboratory tests, as determined by the investigator.
* Has a positive hepatitis panel including anti- hepatitis A virus (only Immunoglobulin M [IgM] is exclusionary), hepatitis B surface antigen, or anti- hepatitis C virus.
* Has a history of human immuno-deficiency virus disease.
* Has a positive urine drug screen including alcohol at Initial Screening or a positive breathalyzer test at any polysomnography check-in.
* Has an apnea hypopnea index (per hour of sleep) >10 (subjects aged 18 to 64) or >15 (subjects aged 65 to 80) as seen on polysomnography, on the first night of the polysomnography screening.
* Has periodic leg movement with arousal index (per hour of sleep) >10 (subjects aged 18 to 64) or >15 (subjects aged 65 to 80) as seen on polysomnography, on the first night of polysomnography screening.
* Has a diastolic blood pressure greater than 90 mm Hg or a systolic pressure of greater than 150 mm Hg.
* The subject has an alanine transaminase level of greater than 3 times the upper limit of normal, active liver disease, or jaundice.
* Has any additional condition(s) that in the Investigator's opinion would:

  * Affect sleep/wake function
  * Prohibit the subject from completing the study
  * Not be in the best interest of the subject.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 472 (Actual)
Dates: Start 2006-07; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Mean wake time after persistent sleep onset during the double-blind Treatment Period, as measured by polysomnography | Weeks 1, 3, and 5 or Final Visit

SECONDARY OUTCOMES:
Number of awakenings after persistent sleep determined by polysomnography. | Weeks 1, 3, and 5 or Final Visit
Latency to Persistent Sleep determined by polysomnography. | Weeks 1, 3, and 5 or Final Visit
Total Sleep Time determined by polysomnography. | Weeks 1, 3, and 5 or Final Visit
Subjective wake time after persistent sleep onset in the sleep lab and at home, as determined by post-sleep questionnaire completed by subject via IVRS. | Weeks 1, 2, 3, 4, and 5 or Final Visit.
Subjective number of awakenings in the sleep lab and at home, as determined by post-sleep questionnaire completed by subject via IVRS. | Weeks 1, 2, 3, 4, and 5 or Final Visit.
Subjective sleep latency using a postsleep questionnaire collected via IVRS. | Weeks 1, 2, 3, 4, and 5 or Final Visit.
Subjective total sleep time using a postsleep questionnaire collected via IVRS. | Weeks 1, 2, 3, 4, and 5 or Final Visit.
Subjective sleep quality using a postsleep questionnaire collected via IVRS. | Weeks 1, 2, 3, 4, and 5 or Final Visit.
Latency to rapid eye movement sleep determined by polysomnography. | Weeks 1, 3, and 5 or Final Visit
Sleep efficiency per polysomnography. | Weeks 1, 3, and 5 or Final Visit

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda

REFERENCES:
- See also: Rozerem Package Insert. — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ROZEREMPI